CLINICAL TRIAL: NCT05971251
Title: Addition of loNcasTuxImab teSirine to AcalabruTinib in Chronic Lymphocytic Leukemia(Anti-Static Study)
Brief Title: Addition of Loncastuximab Tesirine to Acalbrutinib , Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: ADC Therapeutics S.A. (Industry)
Responsible Party: Principal Investigator, Aditi Saha, MD, Assistant Professor, Department of Medicine, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300009213; 000549077 (Other: ADC Therapeutics)
Record Dates: First submitted 2023-07-14; First posted 2023-08-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — loncastuximab tesirine; acalabrutinib

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation based on Dose escalation guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Level 1: (Experimental): 45 µg/kg Loncastuximab Tesirine every 21 days + Acalabrutinib 100 mg BID for 12 cycles
  Interventions: Drug: Loncastuximab Tesirine and Acalabrutinib
- Dose Level 2 (Experimental): 60 µg/kg Loncastuximab Tesirine every 21 days + Acalabrutinib 100 mg BID for 12 cycles
  Interventions: Drug: Loncastuximab Tesirine and Acalabrutinib
- Dose Level 3 (Experimental): 75 µg/kg Loncastuximab Tesirine every 21 days + Acalabrutinib 100 mg BID for 12 cycles
  Interventions: Drug: Loncastuximab Tesirine and Acalabrutinib
- Dose level 4: (Experimental): 90 µg /kg Loncastuximab Tesirine (for first 2 cycles followed by 75µg/kg for subsequent 10 cycles) + Acalabrutinib 100 mg BID for a total of 12 cycles.
  Interventions: Drug: Loncastuximab Tesirine and Acalabrutinib

INTERVENTIONS:
Drug: Loncastuximab Tesirine and Acalabrutinib — Will be given on Day 1 of each cycle with each cycle being 21 days, and is being added to BID Acalabrutinib

SUMMARY:
Study is a phase I study to determine the maximum tolerated dose of adding Loncastuximab Tesirine to Aclabrutinib in the treatment of chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
The study is a phase I study which will employ the Bayesian optimal interval (BOIN) design to find the maximum tolerated dose (MTD).

Approximately 24 Dose-Limiting Toxicity (DLT) evaluable participants will be treated to find MTD with a target DLT rate of 25%, and 4 pre-specified doses. The total number of participants enrolled will depend on the frequency of DLTs and when the MTD is determined. The maximum number of patients at a given dose level is 12.

The dose of acalabrutinib will be fixed and loncastuximab tesirine will be titrated as in dose level table 1 below.

Table 1. Dose levels Dose Level Schedule

1. 45 µg/kg Loncastuximab Tesirine + Acalabrutinib 100 mg BID
2. 60 µg/kg Loncastuximab Tesirine + Acalabrutinib 100 mg BID
3. 75 µg/kg Loncastuximab Tesirine + Acalabrutinib 100 mg BID
4. 90 µg /kg Loncastuximab Tesirine (for first 2 cycles followed by 75µg/kg for subsequent cycles) + Acalabrutinib 100 mg BID

The DLT evaluation period is two cycles (42 days).

Loncastuximab Tesirine will be given as an IV infusion, each cycle is a 21 day cycle, with Loncastuximab Tesirine given day 1 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria For all patients

1. Diagnosis of CLL according to the IwCLL criteria or SLL according to the World Health Organization (WHO) criteria. This includes previous documentation of:

   * Biopsy-proven small lymphocytic lymphoma OR
   * Diagnosis of CLL according to the IWCLL criteria as evidenced by Peripheral blood lymphocyte count of greater than 5 x109/L .
   * Immunophenotype consistent with CLL defined as the predominant population of lymphocytes share both B cell antigens (CD19, CD20 (typically dim expression), or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc).
2. On therapy with acalabrutinib for a minimum of 3 months without evidence of progression as per IWCLL 2018 criteria.
3. Relapsed or Refractory CLL who have received at least one prior therapy before initiation of acalabrutinib
4. Presence of measurable residual disease in the peripheral blood or bone marrow aspirate by NGS based clonoseq test.
5. Adequate organ function as defined below unless attributed to disease involvement:

   * Liver function (bilirubin ≤ 1.5 × ULN, AST and/or ALT <3 x ULN). Patients with Gilbert Disease are permitted irrespective of bilirubin values.
   * Kidney function (crcl > 30ml/min using Cockroft-Gault, based on actual weight).
   * ANC ≥ 1,000/µL, Hgb > 8, Platelet Count ≥ 50,000/ µL. Use of G-CSF is not permitted for up to 7 days prior to enrollment.

Exclusion Criteria:

* Exclusion Criteria For all patients

  1. Current evidence of central nervous system involvement.
  2. Unable to generate clonoseq ID specimen for measurable residual disease tracking.
  3. Completion of an autologous hematopoietic stem cell transplantation within 3 months prior to first dose of study drug.
  4. Prior allogeneic stem cell transplant within 6 months. The patient should not have any active Graft vs. Host disease (GVH) or should be on immune suppressive agents.
  5. Completion of treatment with any radiotherapy, chemotherapy, antibody, immunoconjugates and/or another investigational drug ≤4 weeks (or 5 half-lives of the drug, whichever is shorter) prior to the first dose of study drug. Patients may be enrolled after a minimum of 2 weeks of radiation if radiation was for palliative intent.
  6. Progression of disease on BTK inhibitor.
  7. Unable to tolerate full dose of acalabrutinib at 100 mg twice a day.
  8. Inability to swallow and retain oral medications.
  9. Pregnant women are excluded from this study.
  10. Any active, concurrent, significant illness or disease (other underlying lymphoma) or clinically significant findings including psychiatric and behavioral problems, medical history and/or physical examination findings that would preclude the patient from participation in the study such as:

      * active infection requiring systemic therapy ≤10 days before the first dose of study drug
      * unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association [NYHA] II, III, IV;), myocardial infarction ≤6 months prior to first study drug, uncontrolled cardiac arrhythmia e.g., atrial fibrillation/flutter, cerebrovascular accidents ≤6 months before first dose of study drug
      * Significant (as defined by study doctor) pulmonary disease or disorder
      * any severe or uncontrolled other disease or condition which might increase the risk associated with study participation
  11. Vaccination with live, attenuated vaccines within 28 days prior to the first dose of study medication.
  12. Receiving systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents). The use of inhaled corticosteroids is permitted.
  13. Corticosteroids ≥ 10 mg of prednisone within the last 7 days.
  14. Has had a solid organ transplant within the last 3 years. Note: Patients who have had a Solid organ transplant >3 years ago are eligible if there are no signs/symptoms of graft versus host disease (GvHD) and off immunosuppressive medications as per above.
  15. Known history of hypersensitivity to loncastuximab tesirine
  16. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
  17. Breastfeeding or pregnant
  18. Any other malignancy known to be active, with the exception of

      * Cervical carcinoma of Stage 1A (1A1,1A2) and 1B (1B1,1B2,1B3)
      * Non-invasive basal cell or squamous cell skin carcinoma
      * Non-invasive, superficial bladder cancer
      * Prostate cancer with a current PSA level < 0.1 ng/mL
      * Any curable or localized cancer with a CR of > 2 years' duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 12 months
  Recommended phase 2 dose of loncastuximab tesirine in combination with acalabrutinib

SECONDARY OUTCOMES:
Secondary Objective 1 | 6 months
  undetectable measurable residual disease rate (uMRD) at 6 months of combination therapy in peripheral blood by NGS based clonoseq test
Secondary Objective 2 | 12 months
  Undetectable measurable residual disease rate (uMRD) at 12 months of combination therapy by NGS based clonoseq test.
Secondary Objective 3 | 12 months
  Best Overall response rate (ORR = CR+CRi+PR) of loncastuximab tesirine in combination with acalabrutinib
Secondary Objective 4 | 12 months
  Complete response rate (CRR= CR + CRi) of loncastuximab tesirine in combination with acalabrutinib in achieving a complete response.
Secondary Objective 5 | 12 months
  Progression free survival (PFS) at 12 months after completion of all treatment.
Secondary Objective 6 | 12 months
  Incidence of adverse events (AE) of loncastuximab tesirine in combination with acalabrutinib.
Secondary Objective 7 | 12 months
  Duration of response (DOR) of loncastuximab tesirine in combination with acalabrutinib

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Saha, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No